CLINICAL TRIAL: NCT06013670
Title: Endoscopic Therapy+ β Receptor Blockers and TIPS Preventing Rebleeding in Moderate to High-risk Patients With Liver Cirrhosis, Esophageal and Gastric Varices A Multicenter, Prospective Parallel Open Clinical Study
Brief Title: Standard Therapy and TIPS for Moderate to High-risk Esophageal and Gastric Variceal Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-LCYS-MS-13
Record Dates: First submitted 2023-07-14; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-07

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopy+NSBBs treatment group (Experimental): Endoscopic treatment+NSBBs group: After admission, carvedilol 6.25mg qd p.o. was administered to lower portal vein pressure. After one week without any adverse reactions, add the dosage to 12.5mg qd, maintained for a long time, with close monitoring of blood pressure and pulse (morning and evening monitoring) during dosing and later use, to maintain systolic blood pressure>90mmHg and heart rate>55bpm. Otherwise, dosage reduction or even discontinuation of medication is necessary. Endoscopic treatment adopts sequential treatment, with an interval of four weeks, until the varicose vein becomes mild or disappears.
  Interventions: Procedure: Endoscopy+NSBBs
- TIPS treatment group (Experimental): Patients receives TIPS for the prevention of variceal bleeding
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt

INTERVENTIONS:
Procedure: Endoscopy+NSBBs — Endoscopic treatment+NSBBs group: After admission, carvedilol 6.25mg qd p.o. was administered to lower portal vein pressure. After one week without any adverse reactions, add the dosage to 12.5mg qd, maintained for a long time, with close monitoring of blood pressure and pulse (morning and evening monitoring) during dosing and later use, to maintain systolic blood pressure>90mmHg and heart rate>55bpm. Otherwise, dosage reduction or even discontinuation of medication is necessary. Endoscopic treatment adopts sequential treatment, with an interval of four weeks, until the varicose vein becomes mild or disappears.
  Arms: Endoscopy+NSBBs treatment group
Procedure: Transjugular intrahepatic portosystemic shunt — TIPS group: All TIPS procedures are completed by a professional liver disease intervention treatment team.
  Arms: TIPS treatment group

SUMMARY:
Comparison of endoscopic therapy combined with non-selective therapy β Receptor blockers (NSBBs) and TIPS in the treatment of liver cirrhosis

The impact of reducing bleeding on the survival of critically ill patients. To compare the effect of endoscopic therapy combined with NSBBs drugs and TIPS on rebleeding and incidence of Hepatic encephalopathy in patients with moderate risk of liver cirrhosis hemorrhage.

DETAILED DESCRIPTION:
Portal hypertension (PH) is one of the most common and serious adverse consequences of liver cirrhosis. Its complications, including esophageal and gastric variceal bleeding (EGVB), intractable ascites, Hepatorenal syndrome, have become the main cause of death in patients with liver cirrhosis. In patients with compensated cirrhosis, the incidence of varices is 30% -40%, while in patients with decompensated cirrhosis, the incidence of varices is as high as 85%. Varices progress at a rate of 7% -8% annually, with an annual bleeding rate of 10% -15% and a 6-week mortality rate of 15% -25% [1,2]. Within 1-2 years after the first bleeding, approximately 60% of untreated patients experience variceal rebleeding, with a mortality rate of about 30% [4].

In recent years, both domestic and international guidelines have recommended the use of endoscopic ligation in the absence of effective risk stratification measures

(EVL) Joint Non Selective β Receptor blockers (NSBBs) are the preferred treatment for preventing rebleeding in patients with esophageal and gastric variceal bleeding due to cirrhosis (standard treatment), while for those who fail standard treatment (with rebleeding), transjugular intrahepatic portosystemic shunt (TIPS) is used [4]. Although TIPS is significantly superior to standard treatment in the prevention of rebleeding, its complications are relatively more, especially the portal vein blood flow shunt effectively achieved through TIPS, which leads to Hepatic encephalopathy (HE) caused by insufficient liver perfusion and liver failure. More importantly, previous studies have not found that TIPS can improve patient survival. Two RCTs compared TIPS and EVL for secondary prevention of VB, and concluded that TIPS significantly reduced the occurrence of rebleeding without any significant difference in 2-year survival rate. [8,9] This may be due to bias caused by the lack of risk stratification for patients.

The level of portal vein pressure is closely related to the prognosis of patients. Numerous studies have shown that hepatic vein pressure gradient (HVPG) can reflect the severity of portal hypertension, and it is still the "gold standard" for diagnosing portal hypertension. HVPG has been proven to be the best risk stratification tool for portal hypertension. Recently, it has also received more and more attention and has been carried out more and more widely. [3] Although more and more non-invasive methods can be used in daily clinical practice, non-invasive procedures still cannot replace HVPG in decompensated liver cirrhosis patients. [3] HVPG ≥ 10 mmHg is defined as clinical dominant portal Hypotension (CSPH), and variceal bleeding is prone to occur when HVPG ≥ 12 mmHg; In patients with HVPG ≥ 16 mmHg, the mortality rate of acute variceal bleeding increases; HVPG ≥ 20 mmHg has become an effective predictor of early rebleeding in clinical practice. [12] Recent expert consensus indicates that hierarchical treatment of HVPG is a reasonable clinical strategy.

A domestic study in 2015 concluded that risk stratification based on HVPG contributes to the decision of secondary prevention and treatment strategies for esophageal and gastric variceal bleeding in liver cirrhosis. [13] However, the cut-off point of HVPG in risk stratification has not been clearly demonstrated. Based on the value of HVPG, target patients can be classified as high-risk (HVPG>20mmHg), medium risk (16mmHg ≤ HVPG ≤ 20mmHg), and low-risk (HVPG<16mmHg). Previous studies have shown that HVPG>20mmHg is an independent predictor of rebleeding and frequent death. Therefore, TIPS has been widely recognized as the preferred method for preventing rebleeding in high-risk patients [16]. However, there is no consensus on whether to choose TIPS treatment as high-risk patients for moderate to high-risk patients with 16mmHg ≤ HVPG ≤ 20mmHg. In a small study of 49 patients, the survival probability of patients with baseline HVPG below 16 mmHg was significantly higher than that of patients with HVPG above 16 mmHg. [14] In addition, CandidV et al. pointed out that HVPG>16mmHg is one of the predictive factors for treatment failure in the acute bleeding phase of esophageal and gastric variceal bleeding. [15] However, there is currently no research indicating that TIPS can improve the prognosis of patients at moderate risk.

Our research group has completed three retrospective small sample studies in the early stage. For patients with HVPG ≥ 20 mmHg, TIPS has a significant reduction in rebleeding rate and survival benefits compared to standard treatment (propranolol+EVL), consistent with previous studies. [17] For medium to high-risk patients, TIPS significantly reduced the rate of rebleeding compared to EVL+NSBBs during a 2-year follow-up period, but did not show significant benefits in improving survival. [18] In 2021, our research team conducted a single center retrospective study to compare the clinical efficacy of TIPS and EVL+NSBBs based on HVPG related risk stratification for secondary prevention of EGVB in cirrhotic portal hypertension. During a 5-year long-term follow-up, for patients with HVPG ≥ 16mmHg, patients receiving TIPS can obtain significant survival benefits, and the incidence of dominant Hepatic encephalopathy is not higher than that of the standard treatment group.

To further verify the reliability of this conclusion, a multicenter prospective parallel open clinical study is planned to explore the treatment strategy of secondary prevention for medium risk patients with 16mmHg ≤ HVPG ≤ 20mmHg. Endoscopic therapy combined with NSBBs drug therapy and TIPS prevention of rebleeding in medium risk patients with esophageal and gastric variceal bleeding due to cirrhosis is of great clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as liver cirrhosis (based on clinical, laboratory examination, imaging, or liver biopsy), and the disease is caused by viral hepatitis cirrhosis or alcoholic cirrhosis.
* 16mmHg ≤ HVPG ≤ 20mmHg
* Gastroscopy confirms moderate to severe esophageal and gastric varices (EV and GOV1 types) with at least one history of EGVB
* Age 18-80 years old and liver function CTP grading B or C<14 points
* Sign the informed consent form;
* Expected survival time greater than 1 year

Exclusion Criteria:

* Patients with cirrhosis associated with non viral hepatitis or Alcoholic hepatitis Taking NSBBs or other medications to treat portal hypertension within the past 6 weeks
* Contraindication for the use of NSBBs, such as bronchial asthma, Cardiogenic shock, heart block (Ⅱ - Ⅲ degree atrioventricular block), severe or acute heart failure and sinus bradycardia
* Simultaneously taking drugs that affect the metabolism and absorption of NSBBs in the body
* TIPS recanalization treatment due to shunt failure
* Serum total bilirubin>85.5 µ mol/L
* Preoperative evaluation reveals the presence of liver cancer or extrahepatic tumors, severe organ dysfunction, and other factors that affect expected survival disease
* Intractable ascites or hepatorenal syndrome
* Concomitant portal vein cavernous degeneration or severe portal vein system thrombosis
* Women who plan to become pregnant or are already pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | 24 months
  Refer to Baveno VII standard for definition of rebleeding.
Hepatic encephalopathy | 24 months
  The definition and grading of HE refer to the consensus opinion on the diagnosis and treatment of Hepatic encephalopathy in China in 2013. The observation indicators include dominant HE and MHE (OHE). The evaluation of HE is based on the West Haven grading standard. Spontaneous HE is defined as explicit HE that occurs at least once without a clear cause.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Zhang, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Yuzheng Zhuge, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No